CLINICAL TRIAL: NCT07228767
Title: Assessment of Surgeons' Mental Fatigue Based on Operating Time
Acronym: COGNICHIR
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Other Study IDs: CHD25_0013
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Surgical Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgeons from the Digestive Surgery Department at the Vendée Departmental Hospital Center.

SUMMARY:
In May 2023, the French National Authority for Health published a solution for patient safety regarding tunnel vision. This concept, which is uncommon in the medical field, is defined as any situation in which a professional's attention is so focused on a goal that they do not hear or see warning signs that should prompt them to change their approach or even stop before an adverse event associated with care occurs.

To better understand the causes of medical errors, the research will assess surgeons' mental fatigue and the factors associated with it. This fatigue, which occurs after or during prolonged periods of intense cognitive activity, is associated with a temporary inability to maintain optimal cognitive performance. Assessing mental fatigue is crucial in surgeons, as it can directly affect their ability to perform complex procedures and make critical decisions. The aim of this research is to examine the factors that may influence the level of mental fatigue and cognitive load in surgeons during surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Surgeon working in the digestive surgery department at CHD Vendée
* Surgeon capable of understanding the protocol and willing to participate in the research

Exclusion Criteria:

* Surgeon unable to be available for the entire duration of the research

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Surgeons in the Digestive Surgery Department at CHD Vendée
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2025-12-05 (Estimated); Primary Completion 2027-01-05 (Estimated); Study Completion 2027-01-05 (Estimated)

PRIMARY OUTCOMES:
Measurement of surgeons' mental fatigue using visual analog scales from 0 (no fatigue, perfectly clear mind) to 100 (extreme fatigue, inability to maintain concentration). | Before and after surgical procedures during 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Emeric ABET, Principal Investigator — Centre Hospitalier Départemental Vendée
Locations (1):
- Centre Hospitalier Départemental Vendée, La Roche-sur-Yon, France

IPD SHARING:
Plan to Share IPD: No